CLINICAL TRIAL: NCT00068523
Title: Immunomodulation by Ultraviolet B-Irradiation (UVB) to Facilitate Allogeneic Stem Cell Transplantation for Treatment of Hematologic Malignancies
Brief Title: Ultraviolet-B Light Therapy and Allogeneic Stem Cell Transplantation in Treating Patients With Hematologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Omer N. Koc, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICC7Y02
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: refractory multiple myeloma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; blastic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; relapsing chronic myelogenous leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; secondary myelodysplastic syndromes; Philadelphia chromosome negative chronic myelogenous leukemia; chronic idiopathic myelofibrosis; B-cell chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; chronic phase chronic myelogenous leukemia; recurrent adult Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; secondary acute myeloid leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Anemia, Refractory, with Excess of Blasts; Primary Myelofibrosis; Leukemia, Large Granular Lymphocytic; Leukemia, Myeloid, Chronic-Phase; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Antilymphocyte Serum; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Methylprednisolone; Ultraviolet Therapy; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-thymocyte globulin — anti-thymocyte globulin IV over 4 hours on days -2 to -1
Drug: cyclophosphamide — cyclophosphamide IV over 1 hour on days -3 to -2
Drug: cyclosporine — oral cyclosporine on days -1 to 100
Drug: fludarabine phosphate — fludarabine IV over 30 minutes on days -8 to -4
Drug: methylprednisolone — methylprednisolone (oral or IV) on days 5-15
Procedure: UV light therapy — Patients undergo ultraviolet-B (UVB) light therapy every other day between days -10 and -2 for a total of 3 days. Posttransplantation UVB light therapy: Following PBSC transplantation, patients undergo UVB light therapy twice weekly on week 1 (at least 1 day apart) and three times weekly on weeks 2-4.
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation — Allogeneic peripheral blood stem cell (PBSC) transplantation: Patients undergo PBSC transplantation on day 0.

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy. Sometimes the transplanted cells from a donor are rejected by the body's normal cells. Ultraviolet-B light therapy given before and after allogeneic stem cell transplantation may help prevent this from happening.

PURPOSE: Clinical trial to study the effectiveness of combining ultraviolet-B light therapy with allogeneic stem cell transplantation in treating patients who have hematologic malignancies.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of ultraviolet-B light therapy and allogeneic peripheral blood stem cell transplantation in patients with hematologic malignancies by demonstrating 100-day mortality no greater than 15% and 1-year mortality no greater than 40%.
* Determine the frequency of treatment-related toxicity leading to death and frequency of disease relapse resulting in death in patients treated with this regimen.
* Determine the incidence and severity of acute and chronic graft-versus-host disease in patients treated with this regimen.

Secondary

* Determine the rates of donor allogeneic hematologic engraftment in patients treated with this regimen.
* Determine the rate and quality of immune reconstitution in the peripheral blood and the composition of immune cells in the skin before and after transplantation in these patients.
* Determine the event-free and overall survival of patients treated with this regimen.

OUTLINE:

* Preparative regimen: Patients receive fludarabine IV over 30 minutes on days -8 to -4 and cyclophosphamide IV over 1 hour on days -3 to -2. Patients also receive anti-thymocyte globulin IV over 4 hours on days -2 to -1. Patients undergo ultraviolet-B (UVB) light therapy every other day between days -10 and -2 for a total of 3 days.
* Allogeneic peripheral blood stem cell (PBSC) transplantation: Patients undergo PBSC transplantation on day 0.
* Graft-versus-host disease prophylaxis: Patients receive oral cyclosporine on days -1 to 100 and methylprednisolone (oral or IV) on days 5-15.
* Posttransplantation UVB light therapy: Following PBSC transplantation, patients undergo UVB light therapy twice weekly on week 1 (at least 1 day apart) and three times weekly on weeks 2-4.

Donor lymphocyte infusion is performed per institutional guidelines for patients in whom emerging donor chimerism post allogeneic PBSC transplantation is not progressing (consistently below 50% during first 3 months), for whom donor chimerism is receding (to below 25%) despite cessation of cyclosporine, or who relapse within 24 months after allografting.

Patients are followed at least monthly for 3 months and then at 6, 12, 18, and 24 months.

PROJECTED ACCRUAL: A total of 23-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of any of the following hematologic malignancies:

  * Acute myeloid leukemia (AML) meeting any of the following criteria:

    * First complete remission with high-risk karyotype

      * Translocations t(15;17) allowed only if failed first-line induction therapy OR molecular evidence of persistent disease exists
      * Translocations t(8;21) and inv(16) allowed only if failed first-line induction therapy
    * Second or subsequent complete remission
    * Minimal residual disease*
  * Acute lymphoblastic leukemia meeting any of the following criteria:

    * Failed induction therapy and has minimal residual disease* by salvage therapy
    * First complete remission with high-risk karyotype (e.g., t[4;11] or t[9;22])
    * Relapsed disease allowed provided a second or subsequent complete remission or minimal residual disease* is achieved
  * Chronic myelogenous leukemia meeting any of the following criteria:

    * Persistent or relapsed disease after 1 year of imatinib mesylate therapy
    * Accelerated phase or blast crisis

      * Blast crisis allowed after reinduction chemotherapy places disease in chronic phase
  * Myelodysplastic syndromes meeting any of the following criteria:

    * Refractory to medical management
    * Cytogenetic abnormalities predictive of transformation into acute leukemia, including 5q-, 7q-, monosomy 7 and trisomy 8, or evidence of evolution to AML (e.g., refractory anemia with excess blasts (RAEB) or RAEB in transformation)
  * Non-Hodgkin's lymphoma or Hodgkin's lymphoma meeting any of the following criteria:

    * Beyond first complete remission or failed primary induction therapy and demonstrated sensitivity to therapy during the 6 months before transplantation
    * Recurrent disease after autologous stem cell transplantation

      * Must be at least 3 months posttransplantation
    * Cyclin D1+ mantle cell lymphoma allowed after induction therapy and in first remission
  * Multiple myeloma meeting either of the following criteria:

    * Refractory or relapsed disease
    * Residual disease after autologous transplantation
  * Chronic lymphocytic leukemia (CLL) meeting all of the following criteria:

    * Peripheral blood absolute lymphocyte count greater than 5,000/mm^3
    * Small to moderate size lymphocytes and less than 55% pro-lymphocytes, atypical lymphocytes, or lymphoblasts morphologically
    * B-cell or T-cell
  * Myeloproliferative disorders, including myelofibrosis

    * Philadelphia negative
* Availability of a HLA-A, B, and DR identical family donor OR HLA-A, B, and DR genetically matched unrelated donor
* Must meet 1 of the following criteria:

  * At least 55 years of age at time of transplantation
  * Received extensive prior therapy (i.e., more than 1 year of alkylator therapy or more than 2 different prior salvage regimens) or stem cell transplantation with myeloablative conditioning (either autologous or allogeneic)
  * Presenting with comorbid condition (e.g., abnormal cardiac, pulmonary, or renal function and/or prior life-threatening infection) that precludes eligibility for enrollment in allogeneic transplantation protocols with full ablation conditioning
* No active CNS disease NOTE: *Defined as having no circulating blasts, absolute neutrophil count greater than 1,000/mm3 and less than 10% blasts in bone marrow at least 3 weeks after last systemic chemotherapy

PATIENT CHARACTERISTICS:

Age

* See Disease Characteristics
* Over 18

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* ALT/AST no greater than 4 times normal

Renal

* See Disease Characteristics
* Creatinine less than 2.0 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular

* See Disease Characteristics
* Normal cardiac function by echocardiogram or radionuclide scan
* Shortening fraction or ejection fraction at least 40% of normal

Pulmonary

* See Disease Characteristics
* DLCO at least 60%
* FEV_1 greater than 50% of predicted
* Pulse oximetry greater than 85%

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No uncontrolled active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 2 weeks since prior biologic response modifiers, signal transduction inhibitors, or monoclonal antibodies

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior systemic conventional chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Recovered from prior therapy
* No concurrent sun block/sunscreen or any cosmetic that may act as a sunscreen (e.g., lotion with SPF) on the days of scheduled ultraviolet-B light therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-06; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Study the effectiveness of combining ultraviolet-B light therapy with allogeneic stem cell transplantation in treating patients who have hematologic malignancies. | Patients are followed at least monthly for 3 months and then at 6, 12, 18, and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Omer N. Koc, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States